CLINICAL TRIAL: NCT00280202
Title: Detection of Genetic Markers of Lung Cancer Initiation and Progression
Brief Title: Detection of Genetic Markers of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Arjun Pennathur, MD, University of Pittsburgh
Other Study IDs: STUDY19060269; UPCI #99-053 (Other: UPittsburgh Cancer Institute Protocol Review Committee)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Carcinogenesis; Genomic changes leading to malignant phenotypes in NSCLC.; Simultaneous mutagenesis of epithelial cells.; Chromosomal abnormalities/mutations in bronchial tissues.; Detect micrometastases in histologically neg. lymph nodes
MeSH Terms: conditions — Lung Neoplasms; Carcinogenesis; Chromosome Aberrations | interventions — Bronchoalveolar Lavage; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue, and lymph nodes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsy of the major carinal area — Biopsy performed intraoperatively
Procedure: Biopsy of abnormal & suspicious areas of the bronchial tree — Biopsy performed intraoperatively
Procedure: Evaluation of the tumor for DNA mutations — Tumor tissue is banked for future analysis.
Procedure: Bronchoalveolar Lavage (BAL) for cytokine analysis — BAL performed intraoperatively
Procedure: Correlation of flow cytometric & RT PCR for TNM stage — Tissues banked for future correlative studies
Procedure: Analysis of lymph nodes — Tissues banked for future analysis

SUMMARY:
The purpose of this research study is to determine the genetic changes and immunologic changes that are involved in the development and progression of bronchogenic lung cancer.

DETAILED DESCRIPTION:
The multistage theory of carcinogenesis includes the development of multiple activating genetic changes due to exposure to carcinogens, either primarily, or superimposed upon pre-existing mutations in the genome. These changes result in activation of protooncogenes, lack of expression of tumor suppressor genes, or combinations of the above, the sum of which results in malignant transformation. Detailed analyses of chromosomal lesions in bronchogenic lung cancer reveal several recurring abnormalities, including deletions, duplications or polysomy of chromosomes 1, 3, 7 and 20. Aberrations in the short arm of chromosome 3, in particular, are found in many small cell and non-small cell lung cancers, and polysomy 7 is a frequent finding in non-small cell lung cancers. Many of these abnormalities have no identified significance, however the application of current and evolving techniques of molecular biology have revealed specific genomic changes leading to malignant phenotypes in several tumors, for example, the application of polymerase chain reaction amplification techniques has revealed a striking incidence of mutations in the h- and k-ras protooncogenes have been discovered, associated with over-expression of growth factors or receptors, for example epidermal growth factor receptor.

As all epithelial cells are exposed to similar environmental conditions, it seems likely that many cells undergo mutagenesis simultaneously. Clinically, this is frequently apparent, as 10-20% of patients with lung cancer have another epithelial cancer arise, either concurrently, or at some later time in their course. The predisposition for development of second malignancies also affects other epithelial surfaces, for example, there is a strong tendency for patients with cancer of the head and neck to develop a second malignancy (bronchogenic lung cancer) in the aerodigestive tract. Despite decreases in the smoking rate overall in the United States, projections through 2025 indicate that there will still be 100,000 deaths annually from lung cancer and other smoking-associated cancers. Therefore, it would be of great benefit to patients at risk of developing lung cancer to identify these changes prior to the development of invasive malignant lesions. This is particularly true of patients who have already developed a cancer, or in patients with a strong family history who may have occupational (eg., asbestos) or habitual (eg., cigarette smoke) exposure to carcinogens. Identification of cancers in the pre-clinical stage has been attempted previously, for example with screening chest x-rays or sputum cytologies, however, these approaches have not proven to be beneficial, as current detection methods are not sensitive enough to identify early, non-phenotypic changes. The proposal outlined herein is designed to clarify this issue by examining bronchial tissue from patients at risk for development of a second cancer (patients undergoing primary resection for cure of bronchogenic lung cancer) and assessing the biopsy tissue for the presence of chromosomal abnormalities and mutations in the h- and k-ras protooncogenes. These changes may be present for long periods of time in airway epithelial cells prior to the development of overt pathologic changes, and methods to recognize these changes would be useful to assess and follow patients at risk for developing malignancy.

Importance of lymph node status in lung cancer: In patients with non-small cell lung cancer (NSCLC), tumor stage is the strongest determinant of prognosis. Stratification of patients into stages facilitates individual treatment decisions based on the survival statistics of a population. Within these staged populations however, subsets of patients with apparent early disease will still suffer cancer recurrence. This is due to the inability of current staging methods to detect small numbers of disseminated tumor cells (micrometastases) in these patients. Reverse transcription-PCR (RT-PCR) for cancer related messenger RNA's has been shown to detect the presence of micrometastases in histologically negative lymph node specimens, and these findings correlate with poor outcome. Unfortunately, routine clinical application of this technique has been limited by "false positive" results in control tissues and a low specificity for predicting disease recurrence. We have recently shown that quantitative RT-PCR (QRT-PCR) can discriminate between true and false positives, and that this results in an improved ability to predict recurrence. In this proposal we intend to analyze lymph nodes from patients undergoing surgical resection for NSCLC using quantitative RT-PCR. These patients will then be followed for five years to determine tumor recurrence. The goal is to use QRT-PCR to try and identify which patients are at highest risk for disease recurrence and who may therefore benefit from more aggressive therapies.

Specific Aims

1. To obtain and maintain in cell culture 'normal' bronchial epithelial cells (NBECs), tumors, and organoids from patients undergoing resection for treatment of lung carcinoma and mesothelioma.
2. To harvest NBEC and lung tumors for evaluation of genetic abnormalities.
3. To perform molecular analysis including polymerase chain reaction (PCR) amplification, flow cytometry, immunohistochemistry, and gene analysis of material from NBECs, tumors, adjacent and normal lung and blood for evaluation such as mutations in the K-ras and p53 protooncogenes, as well as other candidate genes and pathways such as those involved in epithelial-mesenchymal transition. In addition, we will look for mutations and alterations of expression of Fas, Fas ligand, and FADD, three molecules which mediate programmed cell death and have recently been shown to be expressed on multiple tumor cells including lung cancer.
4. To analyze cytokines present in lavage fluid, tumors, and lung tissues.
5. To produce T cell cultures from cells present in tumor-draining lymph nodes and in tumor tissue. To isolate, numerically expand as well as phenotypically and functionally characterize human tumor-infiltrating lymphocytes (TILs) and tumor cells for the potential development of future cell therapy clinical studies.
6. To analyze intra-pulmonary and mediastinal lymph nodes for expression of tumor related mRNA's (such as carcinoembryonic antigen (CEA), cytokeratin-19, hepatocyte growth factor, gastrin-releasing peptide (GRP) receptor, and the neuromedin-B (NMB) receptor) as potential evidence of micrometastases.
7. To detect metastatic tumor in bone marrow extracted from discarded rib resection material.
8. To analyze biomarkers and circulating tumor DNA (ctDNA) in biological samples and correlate with imaging analysis, and outcomes.
9. To conduct single cell analysis, genomic, proteomic, metabolomic, microbiome, tumor microenvironment, and immunologic research studies on samples collected.

Significance

Several researchers have already established that chromosomal changes occur in a non-random pattern in non-small cell lung cancer. It appears that these changes correlate with specific genetic changes, resulting in the malignant phenotype. Furthermore, a great deal of experimental evidence supports the multistage theory of carcinogenesis, whereby incremental changes in the genome accumulate, resulting in the malignant phenotype. The final product of the accumulated changes is determined by the cell of origin and the number and severity of changes occurring. We hope to establish that early changes (as expressed by karyotypic changes or by particular point mutations) can be identified which would indicate the likelihood of particular patient developing another malignancy. This information could then be applied to clinical situations, for example, to determine the frequency of clinical follow-up by chest x-ray, screening bronchoscopy, or sputum cytology. Furthermore, the information gathered could help identify one or a few genetic changes necessary for transformation, which could then be explored to further define the transformation process.

The presence of malignant cells in lymph nodes is a critical parameter in the staging of lung cancer patients. Assessment of lymph nodes is currently done by histopathology alone. The long-term survival of lung cancer patients who have Stage IB disease (no known lymph node involvement with a tumor greater than 2 cm) is lower than patients who are Stage IA (no known lymph node involvement with a tumor less than 2 cm). Likewise, the survival rates of patients who are judged to be Stage II based on histologically positive level one lymph nodes is often no better than that of higher stage patients who have level two lymph node involvement. These observations suggest that micrometastases are often present in lymph nodes that are not detectable by histological assessment. This proposal will supplement the histopathological examination of lymph nodes with methods that detect occult metastatic cells to determine whether assigning patients to a higher stage more accurately reflects their disease burden. This could affect subsequent treatment and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of lung cancer, lung metastases from a primary site other than lung, mesothelioma or a radiographic lesion highly suspicious for malignancy
* Written informed consent.
* To be scheduled for a biopsy or surgical resection or have already had a biopsy and/or surgical removal of a lung mass

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be selected from investigator's clinic.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 1996-06; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
The odds ratio for the risk of lung cancer associated with molecular markers | No specific time frame

SECONDARY OUTCOMES:
To obtain/maintain in cell culture "normal" bronchial epithelial cells(NBECs), tumors, and organoids from subjects undergoing resection for treatment of lung carcinoma and mesothelioma. | No specific time frame
To harvest NBEC and lung tumors for evaluation of genetic abnormalities; this will be obtained at the time of bronchoscopy and lung resection. | No specific time frame
To perform molecular analysis including PCR amplification, flow cytometry, immunohistochemistry, and gene analysis from NBECs, tumors, adjacent & normal lung, and blood. | No specific time frame
To look for mutations and alterations of expression of Fas, Fas ligand, and FADD, three molecules which mediate programmed cell death and have recently been shown to be expressed on multiple tumor cells including lung cancer. | No specific time frame
To analyze cytokines present in lavage fluid, tumors, and lung tissues. | No specific time frame
To produce T cell cultures from cells present in tumor-draining lymph nodes and in tumor tissue. To isolate, numerically expand as well as phenotypically and functionally characterize human tumor-infiltrating lymphocytes (TILs) and tumor cells. | No specific time frame
To analyze intra-pulmonary and mediastinal lymph nodes for expression of tumor related mRNAs (such as CEA and cytokeratin-19) as potential evidence of micrometastases. | No specific time frame
To detect metastatic tumor in bone marrow extracted from discarded rib resection material which is sometimes removed for access during resection of the lung. | No specific time frame
To analyze biomarkers and circulating tumor DNA (ctDNA) in biological samples and correlate with imaging analysis and outcomes. | No specific time frame
To conduct single cell analysis, genomic, proteomic, metabolomic, microbiome, tumor microenvironment, and immunologic research studies on samples collected. | No specific time frame

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Pennathur, MD, Principal Investigator — Professor (with tenure) of Cardiothoracic Surgery
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided